CLINICAL TRIAL: NCT07232134
Title: Prospective Non-randomized Multicenter Trial: the Efficacy of Therapy in Patients With Acute Myeloid Leukemia and Down Syndrome in Russia
Brief Title: The Efficacy of Therapy in Patients With Acute Myeloid Leukemia and Down Syndrome in Russia
Acronym: AML-DS-2025
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCHPOI- 2025-8
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: AML (Acute Myelogenous Leukemia); Down Syndrome (DS)
Keywords: AML; Acute Myelogenous Leukemia; Down Syndrome; DS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Down Syndrome | interventions — Cytarabine; Idarubicin; Etoposide; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4 chemotherapy blocks: cytarabine/idarubicin/etoposide, cytarabine/idarubicin, high-dose cytarabine (Other)
  Interventions: Drug: 4 chemotherapy blocks: Course 1 AIE (cytarabine/idarubicin/etoposide), Course 2 AI (cytarabine/idarubicin), Course 3 HAD (high-dose cytarabine (1g)/daunorubicin), Course 4 HA (high-dose cytarabine).

INTERVENTIONS:
Drug: 4 chemotherapy blocks: Course 1 AIE (cytarabine/idarubicin/etoposide), Course 2 AI (cytarabine/idarubicin), Course 3 HAD (high-dose cytarabine (1g)/daunorubicin), Course 4 HA (high-dose cytarabine). — 4 chemotherapy blocks: Course 1 AIE (cytarabine/idarubicin/etoposide), Course 2 AI (cytarabine/idarubicin), Course 3 HAD (high-dose cytarabine (1g)/daunorubicin), Course 4 HA (high-dose cytarabine).

SUMMARY:
This prospective non-randomized multicenter trial created based on protocol ML DS 2006 and aimed at standardization of current therapy approaches and creating a national network for diagnostic, treatment and monitoring of children (0-18 years) with AML and Down syndrome in Russia. Based on the results the investigators expect to increase long-term overall and event-free survival in children with AML and DS and reduce the immediate and remote toxicity of chemotherapy by reducing the dose load of chemotherapeutic drugs.

The study protocol therapy for all patients includes four chemotherapy blocks:

Course 1 AIE (cytarabine/idarubicin/etoposide) Course 2 AI (cytarabine/idarubicin) Course 3 HAD (high -dose cytarabine (1g)/daunorubicin) Course 4 HA (high-dose cytarabine) Safety to be monitored based on CTCAE v5.0

DETAILED DESCRIPTION:
This prospective non-randomized multicenter trial created based on protocol ML DS 2006 and aimed at standardization of current therapy approaches and creating a national network for diagnostic, treatment and monitoring of children (0-18 years) with AML and Down syndrome in Russia. Based on the results the investigators expect to increase long-term overall and event-free survival in children with AML and DS and reduce the immediate and remote toxicity of chemotherapy by reducing the dose load of chemotherapeutic drugs.

Patients to be included: Age 0-18 years

* Diagnosis of AML, MDS and presence of Down syndrome (constitutional trisomy 21 and mutation in the GATA1 gene)
* Signed informed consent

Patients not be included:

* Children with Down syndrome and acute lymphoblastic leukemia (ALL)
* Severe comorbidities with contraindications to the treatment according to the protocol
* Pre-treatment >14 days with intensive induction therapy
* Refusal of all therapy or important elements of therapy

NB: Patients with Transient Abnormal Myelopoiesis (TAM) are eligible for enrollment but will be included in the analysis as a separate group.

Patients with M7 AML, trisomy 21 in the tumor clone (without the Down syndrome phenotype) and mutation in the GATA1 gene should be discussed individually with the protocol group to determine the treatment strategy, as patients with M7 AML and trisomy 21 in tumor clone (without the Down syndrome phenotype) are not included in current version of pediatric AML clinical recommendations.

If a patient meets the inclusion criteria, but cannot/should not receive treatment according to the protocol, he/she can be enrolled in the study as a patient under observation. The results of therapy of patients under observation will not be taken into account in the assessment of treatment efficacy.

The study protocol therapy for all patients includes four chemotherapy blocks:

Course 1 AIE (cytarabine/idarubicin/etoposide) Course 2 AI (cytarabine/idarubicin) Course 3 HAD (high-dose cytarabine (1g)/daunorubicin) Course 4 HA (high-dose cytarabine)/ Efficacy parameters include Response rate; event-free survival (EFS); relapse-free survival (RFS); overall survival (OS); treatment-related mortality, myelogram, MRD Safety to be monitored based on CTCAE v5.0 The AML-DS-2025 protocol does not include a maintenance therapy course in order to reduce toxicity and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-18 years
* Diagnosis of AML, MDS and presence of Down syndrome (constitutional trisomy 21 and mutation in the GATA1 gene)
* Signed informed consent

Exclusion Criteria:

* Children with Down syndrome and acute lymphoblastic leukemia (ALL)
* Severe comorbidities with contraindications to the treatment according to the protocol
* Pre-treatment >14 days with intensive induction therapy
* Refusal of all therapy or important elements of therapy

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2030-07-24 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
event-free survival | up to 2 years
  Response rate; event-free survival (EFS)
relapse-free survival (RFS) | up to 2 years
overall survival (OS) | up to 2 years
treatment-related mortality | up to 2 years

SECONDARY OUTCOMES:
CTCAE | up to 2 years
  Number of adverse events by Common Terminology Criteria for Adverse Events (CTCAE) 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- National medical research center of pediatric haematology, oncology and immulogy named after Dmytriy Rogachyov, Moscow, 117198, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No